CLINICAL TRIAL: NCT00366795
Title: Satavaptan in the Prevention of Ascites Recurrence: a Double-blind, Randomised, Parallel-group Comparison of Satavaptan at 5 to 10 mg Daily Versus Placebo in the Absence of Diuretics in Patients With Recurrent Ascites Due to Cirrhosis of the Liver.
Brief Title: Satavaptan for the Prevention of Ascites Recurrence in Patients With Ascites Due to Cirrhosis of the Liver
Acronym: SPARe-2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated due to safety reason.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC6682; EudraCT : 2006-000132-27; LTS10036
Record Dates: First submitted 2006-08-18; First posted 2006-08-21 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-04

CONDITIONS: Ascites; Liver Cirrhosis
MeSH Terms: conditions — Ascites; Liver Cirrhosis | interventions — satavaptan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Satavaptan (Experimental)
  Interventions: Drug: Satavaptan
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Satavaptan — oral administration once daily
  Other Names: SR121463B
  Arms: Satavaptan
Drug: placebo — oral administration once daily
  Arms: Placebo

SUMMARY:
Primary:

To evaluate the efficacy of satavaptan in the absence of concomitant diuretic drugs in reducing the recurrence of ascites.

Secondary:

To evaluate the tolerability and safety of satavaptan in the absence of concomitant diuretic drugs over a 52-week treatment period in patients with cirrhosis of the liver and recurrent ascites.

The one-year double blind placebo controlled period is extended up to 2 years in a long term safety study (PASCCAL-2).

ELIGIBILITY:
Inclusion Criteria:

* Patients with cirrhosis of the liver.
* Patients resistant to the effects of diuretics, intolerant of diuretics or otherwise unsuitable for treatment with diuretics according to the judgement of the investigator.
* Patients with recurrent ascites having undergone both of the following:

  * therapeutic paracentesis for the removal of ascites in the previous 24 hours with the removal of = or > 4 litres of fluid.
  * at least one other therapeutic paracentesis in the previous 3 months.

Exclusion Criteria:

* Patients with an existing functional transjugular intrahepatic portosystemic shunt (TIPS) or other shunt.
* Known hepatocellular carcinoma.
* Patients with ascites of cardiac origin or due to peritoneal infection (e.g. tuberculosis) or peritoneal carcinoma
* Patients previously exposed to satavaptan in the past 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2006-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Number and time of recurrences of therapeutic paracenteses | up to 12 weeks

SECONDARY OUTCOMES:
Time from randomisation to first recurrence of ascites | study period
Increase in ascites | over 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (21):
- Sanofi-Aventis Administrative Office, Malvern, Pennsylvania, United States
- Sanofi-Aventis Administrative Office, San Isidro, Argentina
- Sanofi-Aventis Administrative Office, Macquarie Park, Australia
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Sarajevo, Bosnia and Herzegovina
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Sofia, Bulgaria
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Kuala Lumpur, Malaysia
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Belgrade, Serbia
- Sanofi-Aventis Administrative Office, Singapore, Singapore
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Wong F, Watson H, Gerbes A, Vilstrup H, Badalamenti S, Bernardi M, Gines P; Satavaptan Investigators Group. Satavaptan for the management of ascites in cirrhosis: efficacy and safety across the spectrum of ascites severity. Gut. 2012 Jan;61(1):108-16. doi: 10.1136/gutjnl-2011-300157. Epub 2011 Aug 11. PMID 21836029